CLINICAL TRIAL: NCT06873048
Title: Short-term Study of Myday Sphere and Myday Toric Lenses in Existing Spherical Soft Contact Lenses Wearers With Low Astigmatism (Pacific)
Brief Title: Short-term Study of Two Soft Contact Lenses in Wearers With Low Astigmatism
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision International Limited (CVIL) (Industry)
Collaborators: Centre for Ocular Research & Education, Canada (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CV-24-42
Record Dates: First submitted 2025-03-07; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Astigmatism; Myopia; Hyperopia
MeSH Terms: conditions — Astigmatism; Myopia; Hyperopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Control Contact Lens (stenfilcon A Sphere) (Experimental): All participants will wear Control Contact Lens for one week (Period 1).
  Interventions: Device: Control Contact Lens (stenfilcon A Sphere)
- Test Contact Lens (stenfilcon A Toric) (Experimental): All participants will wear Test Contact Lens for one week (Period 2).
  Interventions: Device: Test Contact Lens (stenfilcon A Toric)

INTERVENTIONS:
Device: Control Contact Lens (stenfilcon A Sphere) — One week of wear
  Arms: Control Contact Lens (stenfilcon A Sphere)
Device: Test Contact Lens (stenfilcon A Toric) — One week of wear
  Arms: Test Contact Lens (stenfilcon A Toric)

SUMMARY:
The primary objective of the study is to evaluate and compare the performance of two soft contact lens.

DETAILED DESCRIPTION:
The primary objective of the study is to evaluate and compare the performance of two different soft contact lens in existing spherical soft contact lens (CL) wearers with low levels of refractive astigmatism over a 2-week wear period.

ELIGIBILITY:
Inclusion Criteria:

1. At least 17 years and no more than 42 years of age.
2. Have read and signed the study consent form.
3. Are willing and able to follow instructions and maintain the appointment schedule.
4. Are habitual wearer of spherical soft contact lenses (not toric or multifocal design), any brand and any replacement frequency.
5. Are willing to wear the study contact lenses for 6 days a week while in this study and on three days (day 1, Day 7 and Day 13) for at least 12 hours.
6. Are willing to provide a contact email and telephone number and to use a device that allows them to respond to a short online questionnaire every 3 hours on days 1, 7 and 13 of each lens arm, while wearing one of the 2 study lenses.
7. Are non-presbyopic i.e. no requirement for a reading addition for routine daily tasks (self report).
8. Have astigmatism of either -0.50, -0.75, -1.00 or -1.25 DC in each eye by subjective sphero-cylindrical refraction.
9. Achieves at least 0.10 LogMAR in each eye by subjective sphero-cylindrical refraction.
10. Can be fit with available study contact lens powers of between +6.00 to -10.00 DS.
11. Demonstrate an acceptable fit with the study contact lenses.

Exclusion Criteria:

1. Are participating in any concurrent clinical interventional study.
2. Have worn rigid contact lenses in the last 3 months.
3. Have worn soft toric contact lenses in the past 3 months.
4. Have any known active ocular disease or allergies and/or infection.
5. Have clinically significant biomicroscopy findings or have an ocular condition that contraindicate contact lens wear.
6. Have a systemic condition that in the opinion of the investigator may affect a study outcome variable or contraindicate wearing soft contact lenses.
7. Are using any systemic or topical medications that in the opinion of the investigator may affect a study outcome variable or contraindicate wearing soft contact lenses.
8. Have known sensitivity to the diagnostic sodium fluorescein to be used in the study.
9. Have undergone refractive error surgery or intraocular surgery.
10. Are an employee of the Centre for Ocular Research & Education directly involved in this study.

Ages: 17 Years to 42 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-26 (Actual); Primary Completion 2025-08-15 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Contact Lens Comfort | Day 1 (day after dispense), Day 7 and Day 13 at 12 hours contact lens wear
  Contact lens comfort will be measured on the scale of 0-100 where, (0=worst and 100=best)

CONTACTS AND LOCATIONS:
Overall Officials: Lyndon Jones, PhD,FCOptom, Principal Investigator — Centre for Ocular Research and Education
Locations (1):
- School of Optometry & Vision Science, Waterloo, Ontario, Canada